CLINICAL TRIAL: NCT07383766
Title: A Prospective Clinical Study Evaluating the Effects of a Skin Boosting Injectable on the Aesthetic Improvement of Facial Rhytids
Brief Title: Aesthetic Improvement of Facial Rhytids Using Injectables
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erevna Innovations Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EINN-2025-PRENEW-03
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Aesthetic
Keywords: Hydration; Skin Heath; Skin Booster; Hyaluronic Acid; Injectable

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Biweekly Treatment (Active Comparator): Participants randomized to Group 1 : Biweekly Treatment, will undergo three treatments with Revanesse (R) Renew(TM)+ spaced 2 weeks apart.
  Interventions: Device: Revanesse® Renew™+
- Group B: Monthly Treatment (Active Comparator): Participants randomized to Group 2: Monthly Treatment, will undergo three treatments with Revanesse (R) Renew(TM)+ spaced 4 weeks apart.
  Interventions: Device: Revanesse® Renew™+

INTERVENTIONS:
Device: Revanesse® Renew™+ — Revanesse® Renew™+, a sterile, colorless, odorless, transparent, aqueous gel of synthetic origin supplied in pre-filled disposable syringes. Revanesse® Renew™+ is manufactured by Prollenium Medical Technologies Inc. It consists of both low- and high-molecular-weight hyaluronic acid (HA) at a concentration of 14 mg/mL. The product is supplied in pre-filled disposable syringes, each containing 1.2 mL of ready-to-use gel intended for single use.
  The product does not require reconstitution or dilution prior to injection and is administered directly into the superficial to mid-dermal plane according to the manufacturer's instructions.

SUMMARY:
Revanesse® Renew™+ (Prollenium Medical Technologies Inc.) is a non-crosslinked HA skin booster that combines low- and high-molecular-weight HA at a concentration of 14 mg/mL in a sterile aqueous gel for intradermal injection7. This dual-weight formulation provides both rapid hydration and sustained moisture retention, improving dermal suppleness and promoting subtle textural refinement through physiologic hydration rather than volumization.

The present study is designed to compare biweekly and monthly treatment schedules of Revanesse® Renew™+, assessing clinical efficacy, objective biophysical markers, and participant-reported outcomes to inform evidence-based treatment protocols in aesthetic medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to adequately understand the verbal explanations and the written participant information provided in local language and ability and willingness to give consent to participate in the study. Signed and dated informed consent to participate in the study.
2. Participant interested in improving skin quality.
3. Immune-competent adult 30 years of age and older.
4. Has intent to undergo treatment to improve appearance of the facial skin.
5. Willingness to comply with pre-visit instructions, including shaving of facial area (for male participants), to allow for consistent biometric and photographic evaluations.
6. If the participant is a female of childbearing potential, she agrees to use an acceptable form of effective birth control for the duration of the study and is willing to take a urine pregnancy test (UPT) at Baseline and prior to receiving any study treatment.

   Acceptable forms of effective birth control include:
   * Barrier methods of contraception: Condom or occlusive cap (diaphragm or cervical caps) with spermicidal foam/gel/film/ cream/suppository;
   * Bilateral tubal ligation;
   * Combined oral contraceptives (estrogens and progesterone), implanted or injectable contraceptives on a stable dose for at least 28 days prior to Day 1;
   * Hormonal or copper intra uterine device (IUD) inserted at least 28 days prior to Day 1;
   * Vasectomized partner (in monogamous relationship) for at least 3 months prior to screening;
   * Strict abstinence (at least one month prior to Baseline and agrees to continue for the duration of the study or use acceptable form of birth control).
7. Negative UPT for women of childbearing potential at the Baseline visit.
8. Stable lifestyle and skincare regimen for at least 4 weeks

Exclusion Criteria:

1. Known or suspected allergy or hypersensitivity to any components of Revanesse® Renew™+
2. Known allergy or intolerance to topical anesthetics or lidocaine.
3. History of hypersensitivity reactions such as anaphylaxis, angioedema, or other severe allergic responses.
4. History of hypertrophic scarring, keloid formation, or post-inflammatory hyperpigmentation following cosmetic treatments.
5. Tattoos, piercings, or skin bleaching agents in the treatment area that may interfere with assessments, as judged by the Investigator.
6. Previous cosmetic or dermatologic procedures in the treatment area within the following time frames:
7. Previous treatment with cross-linked hyaluronic acid dermal fillers in the treatment area within the last 12 months.
8. Energy-based devices (laser, IPL, RF, ultrasound) in the last 6 months.
9. Microneedling, dermabrasion, mesotherapy, or chemical peels in the last 6 months.
10. Use of topical corticosteroids, retinoids, or depigmenting agents in the treatment area within the past 4 weeks.
11. Current use of immunosuppressive therapy, systemic corticosteroids, or chemotherapy within the last 3 months.
12. History of systemic autoimmune, collagen vascular, or bleeding disorders (e.g., lupus, scleroderma, thrombocytopenia).
13. Current pregnancy, positive urine pregnancy test at screening, breastfeeding, or intent to become pregnant during the study.
14. Participation in another clinical study within the past 30 days or concurrent participation in another interventional trial.
15. Any condition, including psychological, cognitive, or behavioral concerns, that would interfere with the ability to give informed consent, follow the protocol, or comply with follow-up requirements.
16. Initiation of a weight loss program or GLP-1 agonist therapy within 30 days before baseline or planned during study period.
17. Current participation by study personnel, immediate family members, or employees of the Sponsor.
18. History of cancer or previous radiation near or on the area to be treated.
19. Heavy smokers, classified as smoking more than 12 cigarettes per day.
20. Presence of any disease or lesions near or on the area to be treated, e.g.

    1. Inflammation, active or chronic infection in or near the treatment area
    2. Psoriasis, eczema, herpes zoster and acanthosis
    3. Cancer or precancerous condition (e.g. actinic keratosis)
    4. Severe skin laxity, flaccidity, or sagging
    5. Advanced photoaged/ photodamaged skin (e.g., advanced skin elastosis, multiple lentigo solaris lesions) or skin condition (e.g., very crinkled, very thin, fragile skin or severe skin atrophy) in the treatment area that in the Investigator's opinion could interfere with the safety or effectiveness of the study product or injection procedure.
21. Skin coloring/bleaching/tattoo in the treatment area, which, in the Treating Investigator's opinion, would interfere with the study injections and/or study assessment.
22. An underlying known disease, a surgical or medical condition that would expose the participant to undue risk, e.g. history of bleeding disorders, active hepatitis, active autoimmune disease such as connective tissue diseases, systemic lupus erythematosus, polymyositis, dermatomyositis, multiple sclerosis or scleroderma.
23. Use of concomitant medication that have the potential to prolong bleeding times such as anticoagulants or inhibitors of platelet aggregation (e.g., warfarin, clopidogrel, aspirin, baby aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), Omega 3 or Vitamin E), within 14 days prior to injection. Omega 3 and Vitamin E are acceptable only as part of a standard Topical Multivitamin formulation. Cyclooxygenase-2 (COX 2) inhibitors are allowed.
24. Treatment with chemotherapy, immunosuppressive agents, systemic corticosteroids within 3 months before treatment (inhaled or ophthalmic corticosteroids are allowed).
25. Use of hormonal therapy (ex. HRT or contraceptives) unless the participant has been on a stable dose for at least 3 months prior to screening and does not plan to make any changes to the HRT regimen during the study period.
26. Pregnancy (confirmed by positive urine pregnancy test (UPT)/ serum pregnancy test), breast feeding or intends to become pregnant over the duration of the study.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2027-02-25 (Estimated); Study Completion 2027-03-25 (Estimated)

PRIMARY OUTCOMES:
Global Aesthetic Improvement Scale (GAIS) Score Assessed by Blinded Evaluat | Baseline to Week 12 (Group 1) and Week 16 (Group 2)]
  Proportion of participants rated as "improved" (improved, much improved, or very much improved) on the GAIS by a blinded evaluator at the end of the study

SECONDARY OUTCOMES:
Safety and Tolerability of Treatment - Patient reported | Baseline to Week 12 (Group 1) and Week 16 (Group 2)]
  Incidence and frequency of adverse events
Safety and Tolerability of Treatment - Physician recoded | Baseline to Week 12 (Group 1) and Week 16 (Group 2)]
  Incidence and frequency of adverse events
Participant Satisfaction With Treatment | Week 2 to Week 12 (Group 1) and Week 4 to Week 16 (Group 2)
  Proportion of participants who report being at least "satisfied" (satisfied, very much satisfied, or extremely satisfied) on a seven-point participant satisfaction scale Proportion of participants who report being at least "satisfied" (satisfied, very much satisfied, or extremely satisfied) on a seven-point participant satisfaction scale Proportion of participants rated as "improved" (improved, much improved, or very much improved) on the GAIS by a blinded evaluator at the end of the study
Percentage Change in Skin Hydration | Baseline to Week 12 (Group 1) and Week 16 (Group 2)
  The percentage change in skin hydration from baseline to Visit 4,5,6 will be assessed to compare the effects of biweekly versus monthly administration of Revanesse® Renew™+ treatment. Assessment will be made using the Corneometer CM 825 (Courage+Khazaka electronic GmbH).
Change in Transepidermal Water Loss (TEWL) From Baseline | Baseline to Week 12 (Group 1) and Week 16 (Group 2)
  Percentage change in TEWL from Baseline to Visit 4,5,6, measured using the Tewameter TM 21.
Change in Skin Surface Biophysical Parameters From Baseline | Baseline to Week 12 (Group 1) and Week 16 (Group 2)
  Percentage change in surface evaluation of living skin cells (SELS: roughness, scaliness, smoothness, desquamation, and pore size) from baseline to Visit 4,5,6, measured via the VisioScan
Change in Skin Elasticity From Baseline | Baseline to Week 12 (Group 1) and Week 16 (Group 2)
  Percentage change in skin elasticity from baseline to Visit 4,5,6, measured using the Cutometer Dual MPA 580
Change in VISIA® CR Facial Imaging Metrics | Baseline to Week 12 (Group 1) and Week 16 (Group 2)
  Percentage change from Baseline in VISIA® CR-derived facial metrics as assessed by non invasive analysis of facial images

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Nikolis, MD, PhD, Principal Investigator — Erevna Innovations Inc.
Locations (1):
- Erevna Innovations Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No